CLINICAL TRIAL: NCT06817265
Title: Phase III Clinical Study on the Efficacy and Safety of TNTL in the Treatment of Non-proliferative Diabetic Retinopathy(With Syndrome of Yin Deficiency With Internal Heat and Blood Stasis Obstructing the Collaterals of the Eyes)
Brief Title: Clinical Study on the Efficacy and Safety of TNTL in the Treatment of Non-proliferative Diabetic Retinopathy
Acronym: TNTL
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beletalent (Zhuhai) Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TNTL-DR-20241112
Record Dates: First submitted 2025-01-24; First posted 2025-02-10 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-01

CONDITIONS: Non-Proliferative Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNTL Experimental Group (Active Comparator): TNTL, oral, 4 tablets, 3 times a day, after meals. Take it for 24 weeks.
  Interventions: Drug: TNTL
- TNTL Control Group (Placebo Comparator): TNTL simulation preparation，oral, 4 tablets, 3 times a day, after meals. Take it for 24 weeks.
  Interventions: Drug: TNTL simulation preparation

INTERVENTIONS:
Drug: TNTL — oral, 4 tablets, 3 times a day, after meals. Take it for 24 weeks.
  Arms: TNTL Experimental Group
Drug: TNTL simulation preparation — oral, 4 tablets, 3 times a day, after meals. Take it for 24 weeks.
  Arms: TNTL Control Group

SUMMARY:
The goal of this clinical trial is to learn if drug TNTL works to treat non-proliferative diabetic retinopathy in adults. It will also learn about the safety of drug TNTL. The main questions it aims to answer are:

1. Does drug TNTL can improve visual acuity and reduce the degree of retinopathy?
2. What medical problems do participants have when taking drug TNTL? Researchers will compare drug TNTL to a placebo (a look-alike substance that contains no drug) to see if drug TNTL works to treat non-proliferative diabetic retinopathy.

Participants will:

1. Take drug TNTL or a placebo every day for 6 months
2. Visit the clinic once every 4 weeks for checkups and tests
3. Keep a diary of their symptoms and Change from baseline

ELIGIBILITY:
Inclusion Criteria:

* Age range of 18 to 75 years old (including boundary values);
* Conform to the diagnosis of type 2 diabetes and diabetes retinopathy. diabetes retinopathy is classified as NPDR and mild and moderate patients;
* Patients with the best corrected visual acuity (BCVA) of the target eye is ≥ 34 points (ETDRS visual acuity chart, visual acuity equivalent to a score of 20/200, decimal 0.1);
* Patients who meet the syndrome differentiation criteria of Yin deficiency, internal heat, and eye meridian stasis in traditional Chinese medicine;
* During the screening period, glycated hemoglobin (HbA1c) should be ≤ 8.5%;
* Agree to participate in this clinical study and voluntarily sign the informed consent form.

Exclusion Criteria:

* Patients with no light perception in one eye;
* Patients with macular edema who require anti Vascular Endothelial Growth Factor(VEGF) treatment;
* People with other eye diseases, such as retinal artery or vein occlusion, non diabetes retinopathy, retinal detachment, uveitis, glaucoma, corneal ulcer, cataract affecting fundus examination, optic neuropathy and high myopia with fundus changes;
* Patients with acute complications of diabetes (such as diabetes ketoacidosis, hyperglycemia hyperosmolality syndrome, diabetes lactic acidosis, etc.) within one year before the screening period;
* People with other eye related complications of diabetes, such as iris neovascularization, angle neovascularization, and retinal neovascularization;
* acupuncture and moxibustion and other external treatment methods of traditional Chinese medicine were used to treat diabetes retinopathy within one week before enrollment;
* Patients who have used drugs clearly stated in the instruction manual to treat diabetes retinopathy, such as calcium dobesilate, pancreatic kallidinogenase, Qiming Granules, Shuangdan Mingmu Capsules, Compound Danshen Dropping Pills, Tongluo Mingmu Capsules, etc. within 2 weeks before enrollment;
* Patients who have undergone glaucoma, vitreous, retinal and other intraocular surgeries and procedures in the target eye within 3 months before enrollment;
* Patients who have undergone cataract surgery in the target eye within 3 months prior to enrollment and have not yet stabilized according to the researcher's assessment;
* Patients who have received intravitreal injections of anti VEGF antibodies and glucocorticoids in the target eye within 3 months prior to enrollment;
* Patients who have undergone total retinal laser photocoagulation treatment in the target eye;
* For those whose refractive media is turbid and difficult to evaluate fundus images in the target eye;
* Uncontrolled or controlled blood pressure with systolic blood pressure ≥ 160mmHg and/or diastolic blood pressure ≥ 100mmHg;
* When screening, alanine aminotransferase (ALT) or aspartate aminotransferase (AST) should be ≥ 1.5 times the upper limit of normal value;
* Patients with serious kidney disease (such as azotemia and uremia), diabetes foot, etc;
* When screening, individuals with severe primary diseases such as respiratory, cardiovascular, cerebrovascular, endocrine, digestive, and hematopoietic systems, or those with severe mental illnesses should be included;
* Suspected or confirmed history of alcohol or drug abuse;
* Pregnant women, lactating women, or women of childbearing age who are preparing to conceive; Female subjects of childbearing age or male subjects (with partners of childbearing age) who do not agree to voluntarily take effective contraceptive measures within one month after the last dose during the screening period;
* Individuals who are allergic to the drugs or their components used in this experiment;
* Participants who have participated in other clinical trials within the past month;
* The researchers believe that participants should not participate in the clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in best corrected visual acuity (BCVA) from baseline after 24 weeks of medication; | From enrollment to the end of treatment at 24 weeks
  After 24 weeks of medication, the subjects' best corrected visual acuity (BCVA) was checked and compared with the value measured at week 0 to observe the degree of change from baseline value;

SECONDARY OUTCOMES:
Change in best corrected visual acuity (BCVA) from baseline after medication | From enrollment to the end of treatment at 4 weeks,8weeks,12weeks,16weeks,20weeks
  After 4 weeks,8weeks,12weeks,16weeks,20weeks of medication, the subjects' best corrected visual acuity (BCVA) was checked separately and compared with the value measured at week 0 to observe the degree of change from baseline value;
The change and progression rate of ETDRS classification DR Classification from baseline after 12 and 24 weeks of medication; | From enrollment to the end of treatment at 12weeks and 24weeks.
  After 12 weeks，24 weeks of medication, the subjects' ETDRS classification based on the Diabetic Retinopathy Severity Score and compared with the value measured at week 0 to observe the change and progression rate from baseline value as required, with a minimum score of 10 and a maximum score of 90. The higher the score, the more severe it is.
The proportion of subjects whose best corrected visual acuity (BCVA)increased by ≥ 5, ≥ 10, ≥ 15 compared to baseline after medication; | From enrollment to the end of treatment at 4,8,12,16,20, and 24 weeks
  After 4,8,12,16,20,24 weeks of medication, count the proportion of subjects whose best corrected visual acuity(BCVA) increased by ≥ 5, ≥ 10, ≥ 15 compared to baseline
The proportion of subjects whose best corrected visual acuity (BCVA) decreased by ≥ 5, ≥ 10, ≥ 15 compared to baseline after medication | From enrollment to the end of treatment at 4,8,12,16,20, and 24 weeks
  After 4,8,12,16,20,24 weeks of medication, count the proportion of subjects whose best corrected visual acuity(BCVA) decreased by ≥ 5, ≥ 10, ≥ 15 compared to baseline
Changes in fundus condition compared to baseline | From enrollment to the end of treatment at 12 and 24 weeks.
  Changes in fundus condition compared to baseline after 12 and 24 weeks of medication
Changes in retinal macular optical coherence tomography (OCT) compared to baseline | From enrollment to the end of treatment at 12 and 24 weeks.
  Changes in retinal macular optical coherence tomography(OCT) after 12 and 24 weeks of medication compared to baseline
Changes in HemoglobinA1c compared to baseline | From enrollment to the end of treatment at 12 and 24 weeks.
  Changes in HemoglobinA1c levels compared to baseline after 12 and 24 weeks of medication
Changes in fasting blood glucose compared to baseline | From enrollment to the end of treatment at 4,8,12,16,20, and 24 weeks
  Changes in fasting blood glucose levels after 4, 8, 12, 16, 20, and 24 weeks of medication compared to baseline
Effective rate of traditional Chinese medicine syndrome | From enrollment to the end of treatment at 4,8,12,16,20, and 24 weeks
  After medication, use the Traditional Chinese Medicine Syndrome（yin deficiency with internal heat and blood stasis obstructing the collaterals of the eyes） Scale as required to score and calculate the effective rate,the lowest score is 0, the highest score is 30, and the higher the score, the more severe it is.

OTHER OUTCOMES:
Adverse events and reactions | From enrollment to the end of treatment at 24 weeks
  Record adverse events, including number of participants with abnormal vital signs,urine analysis, urinalysis,liver function , etc

CONTACTS AND LOCATIONS:
Overall Officials: Hongsheng Bi, Principal Investigator — Shandong University of Traditional Chinese Medicine Affiliated Eye Hospital
Locations (30):
- China (30):
  - Xuancheng People's Hospital, Xuancheng, Anhui
  - Beijing Chaoyang Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong
  - Shenzhen Eye Hospital, Shenzhen, Guangdong
  - Zhuhai People's Hospital, Zhuhai, Guangdong
  - The First Affiliated Hospital of Guizhou University of Traditional Chinese Medicine, Guiyang, Guizhou
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Shijiazhuang People's Hospital, Shijiazhuang, Hebei
  - Kaifeng Central Hospital, Kaifeng, Henan
  - Luoyang Third People's Hospital, Luoyang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Zhengzhou Second Hospital, Zhengzhou, Henan
  - Taihe Hospital （Affiliated Hospital Of Hubei University Of Medicine）, Shiyan, Hubei
  - Wuhan Puren Hospital, Wuhan, Hubei
  - Yichang Central People's Hospital, Yichang, Hubei
  - The First Affiliated Hospital Of University Of South China, Hengyang, Hunan
  - Wuxi People's Hospital, Wuxi, Jiangsu
  - Affiliated Zhongshan Hospital Dalian University, Dalian, Liaoning
  - Shandong University of Traditional Chinese Medicine Affiliated Eye Hospital, Jinan, Shandong
  - Shandong University of Traditional Chinese Medicine Affiliated Hospital, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Shandong Second Provincial General Hospital, Jinan, Shandong
  - Liaocheng People's Hospital, Liaocheng, Shandong
  - The First People'S Hospitalof Xian Yang, Xianyang, Shanxi
  - Xian No.1 Hospital, Xi’an, Shanxi
  - The First Affiliated Hospital of Xi'an Medical University, Xi’an, Shanxi
  - The Affiliated Hospital of Southwest Medical University, Luzhou, Sichuang
  - Panzhihua Integrated Traditional Chinese and Western Medicine Hospital, Panzhihua, Sichuang
  - Yunnan University Affiliated Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No